CLINICAL TRIAL: NCT03581864
Title: Clinical Outcomes of Implantationof Black Diaphragm Intraocular Lens in Complete Aniridia and Aphakia Due to Posttraumatic Eye Rupture
Status: Completed | Type: Observational
Sponsor: Medical University of Lublin (Other)
Responsible Party: Principal Investigator, Dominika Nowakowska, PhD, Medical University of Lublin
Other Study IDs: 0002
Record Dates: First submitted 2018-05-30; First posted 2018-07-10 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-06

CONDITIONS: Aphakia Due to Trauma; Eye; Rupture, Traumatic, With Loss of Intraocular Tissue; Aniridia
Keywords: aphakia; black diaphragmintraocular lens; eye rupture; aniridia
MeSH Terms: conditions — Rupture; Aniridia; Aphakia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group of 14 patients with post-traumatic complete anirirdia: 14 eyes with post-traumatic complete aniridia and aphakia treated withscleral fixation of BD IOL with measurements included ophthalmological comorbidities, best corrected visual acuity (BCVA), complications, and postoperative interventions.

SUMMARY:
Purpose: To assess long-term outcomes of implantation of black diaphragmintraocular lens (BD IOL) in postraumatic aniridia and aphakia due to eye rupture.

METHODS: This is retrospective consecutive case series of 14 eyes with post-traumatic complete aniridia and aphakia treated withscleral fixation of BD IOL with. Measurements included ophthalmological comorbidities, best corrected visual acuity (BCVA), complications, and postoperative interventions. The average postoperative follow-up period was 36 months.

ELIGIBILITY:
Inclusion Criteria:

post-traumatic complete aniridia and aphakia

Exclusion Criteria:

active ocluar inflammation or infection

Ages: 25 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Best-corrected visual acuity | 10 to 120 months
  The visual acuity measurement with ETDRS chart
The slit lamp examination | 10 to 120 months
  The anterior segment of the eye and eye fundus were examined.
The intrraocular pressure measurement | 10 to 120 months
  The procedure was performed with the Goldman applanation tonometer.
The medical history | 10 to 120 months
  Coexisting eye diseases and post-operative complications were noted.

CONTACTS AND LOCATIONS:
Locations (1):
- General Department of Ophthalmology in Lublin, Lublin, Poland

IPD SHARING:
Plan to Share IPD: No